CLINICAL TRIAL: NCT04141579
Title: Functional Improvement of Non-infarcT relaTed Coronary Artery Stenosis by Extensive LDL-C Reduction With a PCSK9 Antibody
Brief Title: Functional Improvement of Coronary Artery Narrowing by Cholesterol Reduction With a PCSK9 Antibody
Acronym: FITTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL71538.091.19
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Atherosclerosis of Coronary Artery
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Two arms. One treatment arm. One arm with placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Experimental): Evolocumab (140mg) will be administered subcutaneously every two weeks (Q2W) on day 1 through week 12 with personal injectors, containing 1 mL deliverable volume of 140 mg/mL Evolocumab.
  Interventions: Drug: Evolocumab 140 MG/ML [Repatha]
- Comparator arm (Placebo Comparator): Placebo will be administered subcutaneously every two weeks (Q2W) on day 1 through week 12 with personal injectors, containing 1 mL deliverable volume of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML [Repatha] — Evolocumab (also known as Repatha, formerly referred to as AMG 145) is a human monoclonal immunoglobulin G2 (IgG2) that specifically binds to proprotein convertase subtilisin/kexin type 9 (PCSK9) preventing its interaction with the low-density lipoprotein receptor (LDLR). The inhibition of PCSK9 by evolocumab leads to increased LDLR expression and subsequent decreased circulating concentrations of low-density lipoprotein cholesterol (LDL-C).
  Other Names: AMG145; Repatha
  Arms: Treatment arm
Drug: Placebo — Matching placebo
  Other Names: Placebo injection
  Arms: Comparator arm

SUMMARY:
In a large number of patients who experienced an acute coronary syndrome, multiple narrowings of the coronary arteries are identified. Mechanical treatment of the infarct related artery is indisputable, yet mechanical treatment of other bystander lesions in non-infarct related arteries is controversial.

Low-density lipoprotein cholesterol can speed up the formation of these coronary artery narrowings, and can increase the risk of a second event.

The investigators want to investigate if treating patients with the new cholesterol-lowering drug evolocumab in addition to statin therapy ameliorates blood flow and reduces atherosclerotic plaque size compared with placebo. Improved blood flow and a reduction of plaque size could prevent the need for additional stenting or surgery.

DETAILED DESCRIPTION:
In a large number of patients presenting with acute coronary syndrome (ACS) multivessel disease is identified. Mechanical treatment of the infarct related artery (IRA) is indisputable, yet mechanical treatment of other bystander lesions in non-infarct related arteries (non-IRAs) is controversial. Some randomized studies have favored preventive complete revascularization during invasive coronary angiography (ICA) over conservative medical treatment with deferred percutaneous intervention (PCI). Yet patient selection and medical treatment in the conservative medical treatment groups were suboptimal.

Revascularization of lesions in the non-IRA can be guided by fractional flow reserve (FFR). In current practice, a value of 0.80 or lower is often used to mark a functionally significant stenosis at a stabilized moment after initial hyperemic response. However, recent evidence suggests that hyperemic response to adenosine is impaired in patients with ACS, which could underestimate how flow-limiting a non-culprit lesion is as measured by FFR. A large patient-level meta-analysis of multiple FFR trials showed that FFR values below 0.67 most evidently identify those at risk of MI or death. Thus, in patients with values above 0.67, mechanical revascularization has less apparent benefit as compared to patients with values below 0.67. The threshold of 0.67 could be a lower safety margin applied for non-IRA lesions, with percutaneous intervention (PCI) as treatment. For values between 0.67 and 0.85, medical treatment could be optimized using the latest generation LDL-C lowering agents on top of current high-intensity statin therapy (HIST) before directly stenting the lesion.

Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors have shown to induce regression of coronary atherosclerotic plaque volume (PV) in patients with coronary artery disease (CAD). As high-risk lesions with large plaque burden (PB) and lipid content are frequently present in ACS, a rapid response on PB and PV can be expected when starting PCSK9-inhibitors on top of HIST. In addition to plaque size, plaque morphology is important in determining residual risk. Lipid-rich plaques have recently again shown to increase the risk of major adverse cardiac events. Lipid rich plaque can be identified using Near-InfraRed Spectroscopy (NIRS). The amount of lipid is represented in the lipid core burden index (LCBI) and is an independent risk factor for future coronary events. A recent study demonstrated the effect on plaque composition in 52 weeks. In this study, an effect in 12 weeks will be evaluated as a potential independent explanation of reduced events in long-term clinical follow-up studies.The change in plaque volume might be closely related to a change in FFR.

Furthermore, it is now well-appreciated that an ACS, a result of atherosclerotic plaque destabilization, initiates a temporary acceleration of atherogenesis in itself. An ACS induces rapid activation of the bone marrow hematopoietic stem- and progenitor cells resulting in monocytosis and activation of innate immune cells, which subsequently accelerate atherosclerosis progression throughout the body. Hypercholesterolemia also activates the innate immune system bone marrow progenitors resulting in long-term activation of the innate immune system. In patients with familial hypercholesterolemia (FH), PCSK9 treatment reduced monocyte CCR2 expression and ex-vivo migratory capacity. Therefore, in the first weeks after an ACS occurred, there is an optimal time window for preventing atherosclerosis progression by powerful lowering of plasma cholesterol.

This pharmaco-invasive strategy with a combination of HIST and a PCSK9-inhibitor could possibly prevent mechanical revascularization (PCI or CABG) in a large cohort of patients. Evolocumab was the first PCSK9-inhibitor approved for clinical use in 2015 for lowering of LDL-C as an adjunct to diet in patients with FH, primary hypercholesterolemia and in patients with homozygous familial hypercholesterolemia (HoFH). Evolocumab has been evaluated in several large scale studies as GLAGOV (N = 968) and FOURIER (N= 27564) on surrogate and clinical endpoints with important benefits and established safety and tolerability.

In this study we want to investigate the effect of maximal LDL-C reduction by evolocumab in addition to HIST compared to placebo on functional impairment of non-IRA lesions, measured by FFR, and the change in NIRS derived lipid core burden index at the 4mm maximal segment (MaxLCBI4mm) from baseline to follow-up in the non-IRA. Secondly, we want to evaluate the change in multiple plaque characteristics, measured by intravascular ultrasound (IVUS). Finally, we will investigate the change in microvascular function, change in pro-inflammatory monocyte phenotype and explore correlations between on treatment LDL-C, LCBI, plaque characteristics and FFR.

ELIGIBILITY:
Inclusion Criteria (all):

* ACS with PCI of infarct related artery
* MVD
* FFR of non-IRA lesion 0.67 - 0.85
* 18 years old at screening

Exclusion Criteria (any):

Refusal or inability to provide informed consent

* Prior coronary artery bypass graft
* Known left ventricular ejection fraction (LVEF) < 30%
* Untreated functional left main stem stenosis (FFR ≤ 0.80)
* Contra-indication for antithrombotic therapy according to ESC guidelines
* Non-IRA stenosis not amenable for PCI treatment (operator's decision)
* Complicated IRA treatment, with one or more of the following:
* Extravasation
* Permanent no re-flow after IRA treatment (TIMI flow 0-1)
* Inability to implant a stent
* Known severe cardiac valve dysfunction that will require surgery in the follow-up period.
* Severe kidney disease defined as an eGFR < 30 ml/min.
* Known severe liver disease defined as Child-Pugh score of 10-15.
* Female subject is pregnant, breastfeeding or planning to become pregnant or planning to breastfeed during treatment and for an additional 15 weeks after the last dose of investigational product. Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive serum pregnancy test.
* Female subjects of childbearing potential unwilling to use 1 acceptable method of effective contraception during treatment and for an additional 15 weeks after the last dose of investigational product.
* Female subject who has not used an acceptable method(s) of birth control for at least 1 month prior to screening, unless the female subject is sterilized or postmenopausal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Change in FFR from baseline to follow-up in non-IRA lesions. | FFR will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Primary physiological endpoint
Change in lipid core burden index at the 4mm maximal segment (MaxLCBI4mm) from baseline to follow-up of the non-IRA. | LCBI will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Primary imaging endpoint

SECONDARY OUTCOMES:
The change in percent atheroma volume (PAV, %) | IVUS will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Secondary invasive imaging endpoint (measured by IVUS)
The change in normalized total atheroma volume (TAV, mm3) | IVUS will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Secondary invasive imaging endpoint (measured by IVUS)
The change in maximum plaque burden (PB, %) | IVUS will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Secondary invasive imaging endpoint (measured by IVUS)
The change in minimum luminal area (MLA, mm2) | IVUS will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Secondary invasive imaging endpoint (measured by IVUS)

OTHER OUTCOMES:
The correlations between achieved on-treatment LDL-C, the change in FFR, the change in LCBI and the change in PAV | This endpoint is measured at the last study visit (12 weeks)
  Exploratory endpoint
The correlation between baseline NIRS derived MaxLCBI4mm and change in FFR of the non-IRA. | This endpoint is measured at the last study visit (12 weeks)
  Exploratory endpoint
The correlation between change in IVUS-derived plaque characteristics and change in FFR of the non-IRA | This endpoint is measured at the last study visit (12 weeks)
  Exploratory endpoint
Change of microvascular resistance as measured by CFR and IMR | CFR/IMR will be assessed at baseline (0 weeks) and at the last follow-up visit (12 weeks)
  Exploratory endpoint
The correlation between LDL-C reduction and reduction of pro-inflammatory monocyte phenotypes. | Blood for monocyte phenotyping will be drawn at baseline, week 4 and week 12
  Exploratory endpoint
Safety endpoints | This endpoint is measured during the study, and terminates 30 days after the participant received the last dose of study medication.
  Patient-oriented composite endpoint (POCE): composite of all-cause death, any stroke, any MI and any revascularization, unplanned ischemia driven PCI of the target lesion, any unplanned ischemia driven PCI in the total study population. Furthermore, all (serious) adverse events will be listed.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan van Geuns, MD, PhD, Principal Investigator — robertjan.vangeuns@radboudumc.nl
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Mensink FB, Los J, Reda Morsy MM, Oemrawsingh RM, von Birgelen C, Ijsselmuiden AJJ, Meuwissen M, Cheng JM, van Wijk DF, Smits PC, Paradies V, van Wijk DJ, Rai H, Ten Cate TJF, Camaro C, Damman P, van Nunen LX, Dimitriu-Leen AC, van Wely MH, Cetinyurek-Yavuz A, Byrne RA, van Royen N, van Geuns RM. Changes in non-culprit coronary lesions with PCSK9 inhibitors: the randomised, placebo-controlled FITTER trial. EuroIntervention. 2025 Aug 18;21(16):910-920. doi: 10.4244/EIJ-D-24-01065. PMID 40828313
- [Derived] Mensink FB, Los J, Oemrawsingh RM, von Birgelen C, Ijsselmuiden A, Meuwissen M, Cheng JM, van Wijk DF, Smits PC, Paradies V, van der Heijden DJ, Rai H, Ten Cate TJ, Camaro C, Damman P, van Nunen LX, Dimitriu-Leen AC, van Wely MH, Cetinyurek-Yavuz A, Byrne RA, van Royen N, van Geuns RM. Functional and morphological improvement of significant non-culprit coronary artery stenosis by LDL-C reduction with a PCSK9 antibody: Rationale and design of the randomized FITTER trial. Heliyon. 2024 Sep 18;10(19):e38077. doi: 10.1016/j.heliyon.2024.e38077. eCollection 2024 Oct 15. PMID 39430462